CLINICAL TRIAL: NCT07082205
Title: Single-Use Antimalarial Monoclonal Antibodies for Post-Discharge Malaria Prevention in Children With Severe Anaemia or Severe Malaria in Kenya: A Multi-Centre, Parallel-Group, Two-Arm Randomised Placebo-Controlled Non-Inferiority Trial
Brief Title: Monoclonal Antibodies in Children With Severe Anaemia or Severe Malaria to Prevent Malaria After Hospital Discharge
Acronym: L9LS-pd
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSTM REC: 24-020; U01GH002290 (NIH); IAA#AAI24032-001-00000 (Other Grant/Funding Number: National Institute of Allergy and Infectious Diseases, National Institutes of Health (NIAID-NIH))
Record Dates: First submitted 2025-06-24; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Malaria; Severe Malaria; Severe Anaemia; Post Discharge
Keywords: monoclonal antibodies; malaria; post-discharge; prevention; severe anaemia; severe malaria; children
MeSH Terms: conditions — Malaria; Anemia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Experimental Arm: mMAbs Participants will receive the antimalarial monoclonal antibody L9LS Administration: Intravenous (IV) infusion Dosage: 30 mg/kg (calculated with 1 kg weight increments) Schedule: Single dose at enrollment Those in the experimental arm will also receive placebo PDMC treatment instead of standard antimalarial medication, 2 weeks after discharge
  Control Arm: Placebo-mMAbs with Standard PDMC Participants will not receive the L9LS monoclonal antibody but will receive placebo (normal saline) Intravenously.
  PDMC: Will receive three courses of monthly post-discharge malaria chemoprevention following WHO guidelines PDMC Medication: Dihydroartemisinin-piperaquine (DP) PDMC Schedule: Administered at 2, 6, and 10 weeks post-hospital discharge
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimalarial monoclonal antibodies (mMAbs) -L9LS + Placebo-PDMC (Experimental): Participants in the mMAb arm will receive the study agent L9LS IV with a target dose of 30 mg/kg. The IV dose will use 1 kg step increases. They will also receive a course of PDMC-Placebo at 2, 6, and 10 weeks post-discharge
  Interventions: Biological: Antimalarial monoclonal antibodies; Drug: Placebo PDMC
- Placebo-mMAB + Malaria chemoprevention- PDMC (Active Comparator): mMAbs-placebo arm: Participants will receive a single infusion of normal saline and thereafter a course of PDMC with dihydroartemisinin-piperaquine at 2, 6, and 10 weeks post-discharge
  Interventions: Drug: Dihydroartemisinin - Piperaquine (DP); Biological: Placebo mMAB

INTERVENTIONS:
Biological: Antimalarial monoclonal antibodies — L9LS Antimalarial monoclonal antibodies (mMAbs)
  Other Names: L9LS
  Arms: Antimalarial monoclonal antibodies (mMAbs) -L9LS + Placebo-PDMC
Drug: Dihydroartemisinin - Piperaquine (DP) — Post-Discharge Malaria Chemoprevention
  Other Names: PDMC
  Arms: Placebo-mMAB + Malaria chemoprevention- PDMC
Biological: Placebo mMAB — Placebo anti malarial monoclonal antibody (placebo mMAB) which is Normal saline
  Other Names: Normal Saline
  Arms: Placebo-mMAB + Malaria chemoprevention- PDMC
Drug: Placebo PDMC — Placebo PDMC course which comprises placebo DP oral tablets
  Other Names: Placebo DP
  Arms: Antimalarial monoclonal antibodies (mMAbs) -L9LS + Placebo-PDMC

SUMMARY:
Background and rationale: Hospitalised children with severe anaemia remain at high risk of dying or requiring hospital readmission for at least 6 months after discharge. In highly malaria-endemic settings, malaria is a major contributor to these post-discharge readmissions and deaths. In 2022, the World Health Organisation (WHO) recommended post-discharge malaria chemoprevention (PDMC) for children hospitalised with severe anaemia living in malarious areas. Kenya, together with several other countries in sub-Saharan Africa, aims to expand WHO's recommendation and introduce PDMC in children hospitalised with severe anaemia or severe malaria, including children with severe malaria who do not have severe anaemia (e.g. cerebral malaria). PDMC consists of full 3-day treatment courses with long-acting antimalarials given monthly three times after discharge. PDMC is very effective in clinical trials. However, adherence to these monthly 3-day drug treatments is limited under real-life conditions. Furthermore, PDMC provides chemoprevention for about 3.5 months only, while the risk of dying or needing to be readmitted remains high for several more months.

The US National Institutes of Health (NIH) has developed two monoclonal antibodies targeting Plasmodium falciparum malaria (mMAb). These proteins specifically target a highly conserved epitope found on the circumsporozoite protein-1 (CSP-1) of P. falciparum to neutralize it and prevent malaria infection. A key feature of mMAbs is that they can provide protection for up to 6 months with a single dose and thus serve as a "long-acting" drug. Recent placebo-controlled studies in healthy adults in Mali suggest that the first mMAb, CIS43LS, when administered at a dose of 40 mg/kg intravenously (IV), can block 88% of malaria infections for at least 6 months. More recently, studies with a newer mMAb called L9LS, which is anticipated to be more potent than CIS43LS, showed a 74% reduction in uncomplicated clinical malaria by 6 months when administered subcutaneously to healthy Malian children aged 6-10 years by a single subcutaneous (SC) dose of 10-20 mg/kg (NCT05304611). Similar studies with L9LS are ongoing in healthy children under 5 years of age in Siaya, western Kenya (NCT05400655).

Young children admitted to hospitals in highly malaria-endemic areas with severe anaemia or severe malaria are an ideal target group for passive immunoprevention with mMAbs as a single infusion with mMAb while in the hospital could protect this high-risk group during the entire vulnerable post-discharge period.

Overview design: investigators will conduct a 2-arm, multi-centre, individually randomised, placebo-controlled non-inferiority trial in 398 children with severe malaria or severe anaemia. Children will be randomly assigned (1:1) using minimum sufficient balance (MSB) randomisation to receive either mMAb before discharge or 3 courses of monthly PDMC after discharge, according to WHO guidelines. The study will be placebo-controlled. Children in the PDMC arm will receive a placebo infusion with normal saline before discharge; children in the mMAb arm will receive placebo-PDMC. All children will receive standard in-hospital care, including a blood transfusion and treatment for severe malaria where indicated. They will also receive a full 3-day treatment course with the antimalarial artemether-lumefantrine (AL) to clear any existing malaria infections as soon as they have recovered and can take oral medication.

The primary endpoint is the incidence of clinical malaria detected by passive case detection by 6 months post-discharge (the intervention period). Key secondary endpoints include the rates of readmissions and deaths (all children). Children will be followed for another 6 months (post-intervention period) to determine the duration of protection, any long-term impact (e.g., growth) and if mMAbs result in a delayed acquisition of natural protective immunity against clinical malaria Study Interventions: All children will receive standard in-hospital care, including a blood transfusion, antibiotics, and treatment for severe malaria where indicated. All children in both arms will be empirically treated for malaria infection around discharge with a 3-day regimen with artemether-lumefantrine to ensure parasite clearance of any existing parasites. Participants in the mMAb arm will receive the study agent L9LS IV with a target dose of 30 mg/kg. The IV dose will use 1 kg step increases. During the 6-month intervention period, children in the placebo-mMAbs arm will receive three courses of monthly PDMC as per WHO guidelines with dihydroartemisinin-piperaquine (DP) at 2, 6 and 10 weeks post-discharge. Those in the mMAbs arm will receive an identical placebo PDMC

DETAILED DESCRIPTION:
Background and rationale: Hospitalised children with severe anaemia remain at high risk of dying or requiring hospital readmission for at least 6 months after discharge. In highly malaria-endemic settings, malaria is a major contributor to these post-discharge readmissions and deaths. In 2022, the World Health Organisation (WHO) recommended post-discharge malaria chemoprevention (PDMC) for children hospitalised with severe anaemia living in malarious areas. Kenya, together with several other countries in sub-Saharan Africa, aims to expand WHO's recommendation and introduce PDMC in children hospitalised with severe anaemia or severe malaria, including children with severe malaria who do not have severe anaemia (e.g. cerebral malaria). PDMC consists of full 3-day treatment courses with long-acting antimalarials given monthly three times after discharge. PDMC is very effective in clinical trials. However, adherence to these monthly 3-day drug treatments is limited under real-life conditions. Furthermore, PDMC provides chemoprevention for about 3.5 months only, while the risk of dying or needing to be readmitted remains high for several more months.

The US National Institutes of Health (NIH) has developed two monoclonal antibodies targeting Plasmodium falciparum malaria (mMAb). These proteins specifically target a highly conserved epitope found on the circumsporozoite protein-1 (CSP-1) of P. falciparum to neutralize it and prevent malaria infection. A key feature of mMAbs is that they can provide protection for up to 6 months with a single dose and thus serve as a "long-acting" drug. Recent placebo-controlled studies in healthy adults in Mali suggest that the first mMAb, CIS43LS, when administered at a dose of 40 mg/kg intravenously (IV), can block 88% of malaria infections for at least 6 months. More recently, studies with a newer mMAb called L9LS, which is anticipated to be more potent than CIS43LS, showed a 74% reduction in uncomplicated clinical malaria by 6 months when administered subcutaneously to healthy Malian children aged 6-10 years by a single subcutaneous (SC) dose of 10-20 mg/kg (NCT05304611). Similar studies with L9LS are ongoing in healthy children under 5 years of age in Siaya, western Kenya (NCT05400655).

Young children admitted to hospitals in highly malaria-endemic areas with severe anaemia or severe malaria are an ideal target group for passive immunoprevention with mMAbs as a single infusion with mMAb while in the hospital could protect this high-risk group during the entire vulnerable post-discharge period.

Overview design: Investigators will conduct a 2-arm, multi-centre, individually randomised, placebo-controlled non-inferiority trial in 398 children with severe malaria or severe anaemia. Children will be randomly assigned (1:1) using minimum sufficient balance (MSB) randomisation to receive either mMAb before discharge or 3 courses of monthly PDMC after discharge, according to WHO guidelines. The study will be placebo-controlled. Children in the PDMC arm will receive a placebo infusion with normal saline before discharge; children in the mMAb arm will receive placebo-PDMC. All children will receive standard in-hospital care, including a blood transfusion and treatment for severe malaria where indicated. They will also receive a full 3-day treatment course with the antimalarial artemether-lumefantrine (AL) to clear any existing malaria infections as soon as they have recovered and can take oral medication.

The primary endpoint is the incidence of clinical malaria detected by passive case detection by 6 months post-discharge (the intervention period). Key secondary endpoints include the rates of readmissions and deaths (all children). Children will be followed for another 6 months (post-intervention period) to determine the duration of protection, any long-term impact (e.g., growth) and if mMAbs result in a delayed acquisition of natural protective immunity against clinical malaria.

Primary efficacy objective: To assess the efficacy of a single dose of L9LS versus PDMC against microscopy or RDT-confirmed clinical malaria in hospitalised children with severe anaemia or severe malaria by 6 months after investigational product (IP) administration.

Sites: Two hospitals in western Kenya in areas with moderate to intense malaria transmission. The number of hospitals will be expanded if recruitment rates require this.

Study Population: Inclusion criteria: convalescent children aged less than 10 years and weighing ≥5 kg hospitalised with severe anaemia (haemoglobin<5g/dL / Ht<15%) or severe malaria who have become clinically stable and can take or switch to oral medication; post-transfusion Hb >5g/dL, resident in the study area, provision of informed consent by parents or guardian. Exclusion criteria: Children eligible for any of the four doses of the RTS,S or R21 malaria vaccines, HIV-infected or HIV-exposed children on daily cotrimoxazole prophylaxis, blood loss due to trauma, malignancy, known bleeding disorders, known hypersensitivity to study drug, known heart conditions or family history of congenital QT prolongation, or taking medicinal products that are known to prolong the QTc interval, non-resident in the study area, previous participation in the study, known need at enrolment for prohibited medication and scheduled surgery during the 12-month course of the study.

Study Interventions: All children will receive standard in-hospital care, including a blood transfusion, antibiotics, and treatment for severe malaria where indicated. All children in both arms will be empirically treated for malaria infection around discharge with a 3-day regimen with artemether-lumefantrine to ensure parasite clearance of any existing parasites. Participants in the mMAb arm will receive the study agent L9LS IV with a target dose of 30 mg/kg. The IV dose will use 1 kg step increases. During the 6-month intervention period, children in the placebo-mMAbs arm will receive three courses of monthly PDMC as per WHO guidelines with dihydroartemisinin-piperaquine (DP) at 2, 6 and 10 weeks post-discharge. Those in the mMAbs arm will receive an identical placebo PDMC.

Follow-up procedures: Children will be followed for 12 months by passive surveillance (unscheduled sick visits) in 2 phases: a 6-month intervention period to the end of month 6 post-discharge (day 183 inclusive); a 6-month post-intervention period from month 7 to 12 inclusive (day 184 to +1 year minus 1 day following discharge).

Outcome Measures: Primary: Incidence rate of clinical malaria from 3 to 26 weeks post-discharge, defined as an illness accompanied by measured fever ≥37.5°C or a history of fever (subjective or objective) in the previous 24 hours, accompanied by any level of asexual parasitaemia detected by microscopy or RDT (pLDH or HRP2-band). The HRP2-band results will only be considered when microscopy or the RDT pLDH band results are unavailable. Key secondary outcomes include the following outcomes measured during the follow-up periods (intervention and post-intervention): All-cause and cause-specific readmissions, all-cause non-severe sick-child clinic visits and those unrelated to malaria, and the pharmacokinetic parameters of L9LS. Other secondary efficacy outcomes include those measured during cross-sectional surveys conducted at the end of the intervention and post-intervention periods, including the prevalence of malaria infection, clinical malaria, anaemia, and standard anthropometric measures of malnutrition. Exploratory endpoints include immunological endpoints. Safety endpoints include solicited and unsolicited AEs (local and systemic) following mMAb administration and anti-drug antibodies (ADA) at 6 and 12 months.

Sample size: This will be a parallel, 2-arm, placebo-controlled, non-inferiority trial using a 1:1 allocation ratio. In this non-inferiority trial, investigators will compare mMAbs against monthly PDMC, assuming higher incidence rates are worse. The primary endpoint is clinical malaria during 24 weeks between 3 and 26 weeks post-discharge. The non-inferiority ratio is 1.1. To demonstrate non-inferiority with 90% power and a one-sided significance level of 0.025 and assuming a potential reduction by mMAbs relative to PDMC of 54% (IRR=0.456) from 72 to 33 per 100 person-years, the study requires approximately 398 participants (199 per arm), considering a 15% dropout rate and an overdispersion parameter of 1.18. The trial includes two interim analyses for efficacy and sample size re-estimation when 50% and 75% of participants have completed their 6-month follow-up.

Data Analysis: The primary analysis will use the modified intention-to-treat population, including all randomised participants contributing to the outcome. Incidence rates will be calculated, and incidence rate ratios will be estimated using negative binomial regression by treatment as randomised. The analysis time will be divided into a) the intervention period (first 6 months, primary analysis), b) the post-intervention period (6-12 months), c) and the cumulative effect by 12 months. If non-inferiority is demonstrated, an analysis for superiority will be conducted.

Impact: The potential application of mMAb would be routine administration to hospitalised children with severe anaemia or severe malaria in highly malarious areas. The potential benefits include the prevention of post-discharge deaths, readmissions, and malaria episodes in these vulnerable groups of children.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for enrolment into the pre-study screening period

* Aged <10 years of both sexes
* Severe anaemia or severe malaria: Initially hospitalised with haemoglobin <5.0 g/dl or PCV <15%, or requirement for blood transfusion for other clinical reasons on or during admission to the hospital, or severe malaria, defined as a requirement for parenteral artesunate in the opinion of the treating clinician and the presence of microscopy or RDT confirmed Plasmodium infection
* Resident in catchment area

Eligibility criteria for enrolment

* Fulfilled the pre-study screening eligibility criteria
* Post-transfusion haemoglobin >=5.0 g/dl or PCV >=15%
* Clinically stable, able to take oral medication, able to feed (for breastfeeding children) or eat (for older children) and able to sit unaided (for older children who were already able to do so before hospitalisation)
* Provision of informed consent by parent or guardian Exclusion criteria for enrolment into the pre-study screening period

Exclusion Criteria:

Exclusion criteria for enrolment into the pre-study screening period

* Recognised specific other causes of severe anaemia (i.e., trauma, haematological malignancy, known bleeding disorders, such as haemophilia)
* Sickle cell anaemia/sickle cell disease
* Body weight <5 kg
* HIV infection or on daily cotrimoxazole prophylaxis

Exclusion criteria for enrolment

* Previous enrolment in the present study
* Children who are scheduled to receive any of the four doses of the malaria vaccine within 6 months after enrolment.
* Received any RTS,S or R21 malaria vaccine primary series or booster dose within the last 14 days inclusive
* On or eligible for cotrimoxazole prophylaxis for HIV infection or HIV exposure
* Children with sickle cell disease because they are eligible for daily proguanil
* Known hypersensitivity to artemether-lumefantrine or dihydroartemisinin-piperaquine
* Anticipated to reside for more than 1 month of the 6-month (26 weeks) intervention period outside of the catchment area (e.g. boarding school)
* Use or known need at enrolment for concomitant prohibited medication during the first 6 months post-discharge
* Ongoing or planned participation in another clinical trial involving ongoing or scheduled treatment with prohibited medicinal products or active follow-up during the first 26 weeks post-discharge
* A known need at the time of enrolment for scheduled surgery during the first 6 months post-discharge
* Suspected non-compliance with the follow-up schedule and protocol in the opinion of the investigator
* Known heart conditions or family history of congenital prolongation of the QTc interval, or taking medicinal products that are known to prolong the QTc interval

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 398 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of clinical malaria from 3 to 26 weeks post-discharge | 3 to 26 weeks post-discharge
  Assess the efficacy of a single dose of L9LS versus PDMC against microscopy or RDT-confirmed clinical malaria in hospitalised children with severe anaemia or severe malaria. Clinical malaria defined as an illness accompanied by measured fever ≥37.5°C or a history of fever (subjective or objective) in the previous 24 hours, accompanied by any level of asexual parasitaemia detected by microscopy or RDT (pLDH or HRP2-band).

SECONDARY OUTCOMES:
Number of participants with adverse events following a dose of L9LS versus PDMC in children hospitalised with severe anaemia or severe malaria | From enrollment to12 months post-discharge
  Assess the safety and tolerability of a single dose of L9LS versus PDMC in children hospitalised with severe anaemia or severe malaria through number of participants with solicited and unsolicited adverse events following intervention product administration.
Efficacy of a single dose of L9LS versus PDMC against the first or only microscopy or RDT-confirmed clinical malaria in children hospitalised with severe anaemia or severe malaria by 6 months post-discharge | 3-26 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against the first or only microscopy or RDT-confirmed clinical malaria in children hospitalised with severe anaemia or severe malaria by 6 months post-discharge. the end point includes the first or only episode of clinical malaria from 3 to 26 weeks post-discharge, inclusive, by time-to-event analysis.
Efficacy of a single dose of L9LS versus PDMC against clinical malaria with parasite density >5,000/microlitre (3- 26 weeks post discharge) | 3-26 weeks post discharge (6 months)
  To assess the efficacy of a single dose of L9LS versus PDMC against clinical malaria with parasite density >5,000/microlitre (3-26 weeks post-discharge)
Efficacy of a single dose of L9LS versus PDMC against readmission for any reason in children hospitalised with severe anaemia or severe malaria by 6 months post-discharge | 3-26 weeks post-discharge (6 months)
  To assess the efficacy of a single dose of L9LS versus PDMC against re-admission from any cause.
Efficacy of a single dose of L9LS versus PDMC on anaemia by 6 months post-discharge | 6 months post discharge
  To assess the efficacy of a single dose of L9LS versus PDMC on Hb and anaemia by 6 months post-discharge. The end points include: Mean Hb at 6 months, Prevalence of any anaemia (Hb<11 g/dL), mild anaemia (Hb 10.0-10.99 g/dl), moderate anaemia (Hb 7.0-9.99 g/dL) and moderate-severe anaemia (Hb<7.0 g/dL) at 6 months
The incidence of clinical malaria from 27 to 52 weeks post-discharge | 27 - 52 weeks post discharge (post intervention)
  To assess the efficacy of L9LS vs PDMC on incidence of clinical malaria from 27-52 weeks post-discharge,
The prevalence of malaria infection and parasite densities at 12 months | 12 months post discharge
  To assess whether protection by a single dose of L9LS versus PDMC in children hospitalised with severe anaemia or severe malaria results in delayed malaria after the effect of L9LS has waned. The end-points is the prevalence of malaria infection and parasite densities at 12 months.
Prevalence of mild (Z-score <-2) and severe (Z-score <-3) of low MUAC-for-age, low weight-for-age, low height-for-age, and low height-for-weight at 12 months | 12 months
  To assess the efficacy of a single dose of L9LS versus PDMC on physical growth by 12 months post-discharge, this involves mean Z scores and prevalence of mild (Z-score <-2) and severe (Z-score <-3) of low MUAC-for-age, low weight-for-age, low height-for-age, and low height-for-weight at 12 months (using the WHO child growth standards).
Efficacy of a single dose of L9LS versus PDMC against cause-specific readmissions (3-36 weeks post-discharge) | 3-26 weeks post discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against cause-specific readmissions (severe malaria, severe anaemia, severe malarial anaemia, severe non-malarial anaemia, readmissions for severe malaria or severe anaemia [composite], readmission for other reasons) (3-26 weeks post-discharge)
Death from any cause (3-26 weeks post discharge) | 3-26 weeks post discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against death from any cause (by 6 months , 3-26 weeks post discharge)
To assess the efficacy of a single dose of L9LS versus PDMC on growth by 6 months post discharge | 6 months post discharge
  Assess the mean Z-scores for mid-upper arm circumference (MUAC) for-age, weight-for-age, height-for-age, and height-for-weight (using the WHO child growth standards) in children who received L9LS versus PDMC at 6 months. Weight will be measured in Kilograms and height in centimeters. these measurements will be converted to Z-scores.
Prevalence of malaria infection detected by microscopy, RDT or PCR at 6 months | 6 months
  Prevalence of malaria infection detected by microscopy, RDT or PCR (composite, microscopy, RDT any band, PCR) at 6 months
Prevalence of malaria infection detected by microscopy, RDT or PCR at 12 months | 12 months
  Prevalence of malaria infection detected by microscopy, RDT or PCR (composite, microscopy, RDT any band, PCR) at 12 months
Sick-child clinic visits for any reason (all-cause) (3-26 weeks post-discharge) | 3-26 weeks post discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits for any reason (all-cause) (3-26 weeks post-discharge)
Sick-child clinic visits unrelated to malaria (all-cause minus primary outcome) (3-26 weeks post-discharge) | 6 months
  To assess the efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits unrelated to malaria in children hospitalised with severe anaemia or severe malaria by 6 months post-discharge
Efficacy of a single dose of L9LS versus PDMC against readmission or death from any cause (composite) (3-26 weeks post-discharge). | 3-26 weeks post discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against readmission or death from any cause (composite) (3-26 weeks post-discharge).
Efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits for any reason (all-cause) (27-52 weeks post-discharge) | 27-52 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits for any reason (all-cause) (27-52 weeks post-discharge)
Efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits unrelated to malaria in children hospitalised with severe anaemia or severe malaria by 12 months post-discharge | 27-52 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against sick-child clinic visits unrelated to malaria in children hospitalised with severe anaemia or severe malaria by 12 months post-discharge
Efficacy of a single dose of L9LS versus PDMC against readmission or death from any cause (composite) (27-52 weeks post-discharge) | 27-52 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against readmission or death from any cause (composite) (27-52 weeks post-discharge)
Death from any cause (27-52 weeks post discharge) | 27-52 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against death from any cause (by12months , 27-52 weeks post discharge)
Efficacy of a single dose of L9LS versus PDMC against cause-specific readmissions (27-52 weeks post-discharge) | 27-52 weeks post-discharge
  To assess the efficacy of a single dose of L9LS versus PDMC against cause-specific readmissions (severe malaria, severe anaemia, severe malarial anaemia, severe non-malarial anaemia, readmissions for severe malaria or severe anaemia [composite], readmission for other reasons) (27-52 weeks post-discharge)

OTHER OUTCOMES:
The maximal observed blood concentration (Cmax) of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria | over 12 months post-discharge
  The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria. This includes the pharmacokinetic parameters of antibody concentration Maximal observed blood concentration (Cmax)
Effect of a single dose of L9LS versus PDMC on biomarkers of inflammation post-discharge in children hospitalised with severe anaemia or severe malaria | Over 12 months post-discharge
  To assess the effect of a single dose of L9LS versus PDMC on biomarkers of inflammation post-discharge in children hospitalised with severe anaemia or severe malaria by Inflammatory biomarkers, such as alpha-1-acid glycoprotein (AGP) and C-reactive protein (CRP).
Effect of a single dose of L9LS versus PDMC on biomarkers of naturally acquired immunity post-discharge in children hospitalised with severe anaemia or severe malaria | Over 12 months post-discharge
  To asses the effect of a single dose of L9LS versus PDMC on biomarkers of naturally acquired immunity post-discharge in children hospitalised with severe anaemia or severe malaria. This will be by IgG responses to blood-stage antigens, such as antibodies to merozoite antigens, including AMA1, MSP1
Intervention costs and costs of health consequences of a single dose of post-discharge L9LS versus PDMC in children hospitalised with severe anaemia or malaria, and their caregivers' willingness to pay for it. | over 12 months post- discharge
  To determine the intervention costs and costs of health consequences of a single dose of post-discharge L9LS versus PDMC in children hospitalised with severe anaemia or malaria, and their caregivers' willingness to pay for it. this entails Costs of intervention, including costs of health consequences, that covers, Provider and patient (household) costs associated with routinely providing MmABs or PDMC and, Provider and patient (household) costs associated with primary admission and readmission or clinic visits of participating children during the follow-up period.
  Caregivers' willingness to pay-estimate
The pharmacokinetic parameters of antibody concentration: Total AUC from Time=0 to the last measurable L9LS concentration and partial AUCs | over 12 months
  The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria. This includes the pharmacokinetic parameters of antibody concentration- Total AUC from Time=0 to the last measurable L9LS concentration and partial AUCs
The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria- Time-weighted average concentrations (Cave) | over 12 months pos-dose
  The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria. This includes- time-weighted average concentrations (Cave)
The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria- Blood terminal elimination rate constant (λz) | over 12 months
  The pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria. This includes Blood terminal elimination rate constant (λz)
Pharmacokinetics of antibody concentrations of a single dose of L9LS in children hospitalised with severe anaemia or severe malaria-AUC from Time=0 extrapolated to infinity (AUC 0-infinity) | over 12 months
  Pharmacokinetic parameters of antibody concentration, including AUC from Time=0 extrapolated to infinity
Pharmacokinetic parameters of antibody concentration- AUC post-final PK collection | 12 months
  AUC post-final PK collection (AUC last-infinity)
Pharmacokinetic parameters of antibody concentration- Clearance (CL), central and peripheral volumes of distribution (Vd1 and Vd2), volume of distribution at steady-state (Vdss), and intercompartmental clearance (Q) | 12 months
  Pharmacokinetic parameters of antibody concentration that includes Clearance (CL), central and peripheral volumes of distribution (Vd1 and Vd2), volume of distribution at steady-state (Vdss), and intercompartmental clearance (Q)
Pharmacokinetic parameters of antibody concentration-Alpha and Beta half-lives | 12 months
  Pharmacokinetic parameters of antibody concentration- Alpha and Beta half-lives

CONTACTS AND LOCATIONS:
Overall Officials: Feiko O Ter Kuile, MD, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (2):
- Kenya (2):
  - HomaBay County Teaching and Referral Hospital, Kisumu, Nyanza
  - Siaya County Referral Hospital, Kisumu, Nyanza

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data will be made available for any individual-participant data meta-analyses, with the understanding that the results of the meta-analysis will not be published before the results of the individual trial without the prior agreement of the investigators. No later than 3 months after the publication of the trial, a fully de-identified data set will be available for sharing purposes.
Supporting Information: Study Protocol
Time Frame: No later than 3 months after the publication of the trial
Access Criteria: Before publication, a request to the investigators will be required and completion of data sharing request will be needed. After publication, any interested professional will have access to the data that will be made available